CLINICAL TRIAL: NCT06182345
Title: Spray Skin Treats in the Treatment of Pediatric Burns
Brief Title: Spray Skin Treats for Pediatric Burns
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hu Zhicheng, Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: SYSU-FAH-20231208
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Burn
Keywords: Pediatric burn; Spray skin; skin graft
MeSH Terms: interventions — Skin Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experiment gourp: Autologous skin cell suspension combined with autologous skin graft was used to treat burn wound
  Interventions: Procedure: spray skin
- Control group: Autologous skin graft was used to treat burn wound
  Interventions: Procedure: skin graft

INTERVENTIONS:
Procedure: spray skin — autologous skin cell suspension combined with skin graft
  Groups: Experiment gourp
Procedure: skin graft — skin graft
  Groups: Control group

SUMMARY:
The treatment of burns in children remains a global challenge. At present, the clinical treatment plan is still waiting for further improvement. This study intends to retrospectively analyze the experience of treating children burn in recent years and promote sharing and application.

DETAILED DESCRIPTION:
The treatment of burns in children remains a global challenge. Children's burn wounds have many characteristics that are different from those of adults, such as easy deepening of the wound, uncooperation in dressing change, poor resistance and so on. At present, there are new dressing applications a nd surgery in clinical treatment, etc., but how to treat children to achieve better therapeutic effects still needs to be explored. This study intends to retrospectively analyze the experience of treating children burn in recent years and promote sharing and application.

ELIGIBILITY:
Inclusion Criteria:

* burn for any reasons
* Children

Exclusion Criteria:

* Combined with mental illness
* Congenital immune disease
* Severe cardiopulmonary failure，etc

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with burns from various reasons
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
take rate | postoperative day 4 weeks
  take rate of skin graft

SECONDARY OUTCOMES:
complication rate | through study completion, an average of 6 months
  after skin grafting, skin infection, necrosis, subcutaneous hematoma, etc

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Zhu, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Department of Burn Surgery, The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No